CLINICAL TRIAL: NCT00567866
Title: Methamphetamine-Quetiapine Interaction in Humans: A Pilot Study
Brief Title: Methamphetamine-Quetiapine Interactions in Humans
Status: Terminated | Phase: Early Phase 1 | Type: Interventional
Why Stopped: Study was terminated due to insufficient funds
Sponsor: University of Arkansas (Other)
Responsible Party: Carole Hamon, University of Arkansas for Medical Sciences
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: 72900
Record Dates: First submitted 2007-12-03; First posted 2007-12-05 (Estimated); Last update posted 2010-07-13 (Estimated); Status verified 2010-07

CONDITIONS: Methamphetamine Dependence
MeSH Terms: interventions — Quetiapine Fumarate

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 1 (Experimental): placebo -50 mg quetiapine- 100 mg quetiapine
  Interventions: Drug: Quetiapine
- 2 (Experimental): 50 mg quetiapine -100 mg quetiapine- placebo
  Interventions: Drug: Quetiapine
- 3 (Experimental): 50 mg quetiapine -placebo- 100 mg quetiapine
  Interventions: Drug: Quetiapine

INTERVENTIONS:
Drug: Quetiapine — 50 or 100 mg of quetiapine orally

SUMMARY:
This study will test the ability of a medicine (Quetiapine) that is used to treat schizophrenia or bipolar disorder to reduce the effects of methamphetamine that make it difficult for users to stop using it. This study will test the ability of a medicine that is used to treat schizophrenia or bipolar disorder to reduce the effects of methamphetamine that make it difficult for users to stop using it. The investigator thinks quetiapine will lessen the effects of methamphetamine.

DETAILED DESCRIPTION:
The specific goal of this project is to examine whether quetiapine will alter the behavioral effects of methamphetamine without producing major cardiovascular changes or toxic effects under controlled laboratory conditions. This goal will be accomplished using a methamphetamine challenge procedure in which quetiapine will be given orally prior to intravenous (iv) methamphetamine administration. This will allow rapid and systematic evaluation of the therapeutic potential of this medication.

Results of this drug-interaction study will help determine further investigations of the clinical efficacy of this and other dopamine-active agents. We hypothesize that quetiapine will reduce the self-reported, performance and cardiovascular effects of methamphetamine.

ELIGIBILITY:
Inclusion Criteria:

1. Must be between the ages of 18-50.
2. Must have experience with IV methamphetamine use, with self-reported recent history of weekly use being greater than the total administered in the study. Recent use will be confirmed by a urine toxicology screen positive for amphetamines. We will recruit moderate to frequent users of methamphetamine. Moderate use is defined as use from once or twice every six weeks to weekly. Frequent users are defined as individuals who use greater than weekly.
3. Must have recent use confirmed by a urine toxicology screen positive for amphetamines.
4. Must not be seeking treatment for methamphetamine abuse/dependence.

Exclusion Criteria:

1. Ill health (major cardiovascular, renal, endocrine, hepatic disorder).
2. Current diagnosis of other drug or alcohol physical dependence (other than nicotine or caffeine).
3. History of major organic psychiatric disorder (psychosis, schizophrenia, bipolar, mania) or significant psychiatric symptoms at the time of evaluation for study participation, including suicidal ideation.
4. Pregnancy, plans to become pregnant or fertile women without adequate means of contraception.
5. Present or recent use of over-the-counter or prescription psychoactive drug or drugs that would have major interaction with drugs to be tested.
6. Medical contraindication to or prior serious adverse effects from methamphetamine or stimulants (i.e., seizures, cardiac arrest) or medical contraindication to test agents (see risks section). Significant physical or psychiatric illness which might impair the ability to safely complete the study or that might be complicated by the study drugs, including prior seizures (after age 8) or other active neurological disease or clinically significant abnormalities on physical examination or screening laboratory values.
7. Current enrollment in a methamphetamine, alcohol, or other drug treatment program or current legal problems relating to methamphetamine, alcohol, or other drug use, including awaiting trial or supervision by a parole or probation officer
8. Body Mass Index >30 or <18
9. Currently trying to quit methamphetamine use or seeking treatment for methamphetamine use
10. History of serious adverse event or hypersensitivity to methamphetamine or other study drugs
11. Currently taking any medication (including highly active antiretroviral therapy (HAART) for HIV) other than over-the-counter nonsteroidal anti-inflammatory medications, topical medications, inhaled asthma therapy, and over-the-counter nonsedating antihistamines
12. Use within the last month of the Vicks Nasal Inhaler or medications that are metabolized to methamphetamine (e.g. selegiline)

    -

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2008-01; Primary Completion 2009-09 (Actual); Study Completion 2009-09 (Actual)

PRIMARY OUTCOMES:
Behavioral Responses to Methamphetamine following predosing with placebo or test article. | Prior to drug administration, and 10 minutes post-drug administration and then hourly for 9 hours

SECONDARY OUTCOMES:
Physiological Responses to methamphetamine following predosing of placebo or test article | Pre-drug dosing, 5, 20, 35, and 50 minutes postdosing until 4 hours postodose, and then twice hourly until the seventh hour

CONTACTS AND LOCATIONS:
Overall Officials: William Brooks Gentry, MD, Principal Investigator — University of Arkansas
Locations (1):
- University of Arkansas for Medical Sciences, Little Rock, Arkansas, United States